CLINICAL TRIAL: NCT03269994
Title: A Phase III Multicenter, Open Label Randomized Controlled Trial of Cefoxitin Versus Piperacillin-Tazobactam as Surgical Antibiotic Prophylaxis in Patients Undergoing Pancreatoduodenectomy
Brief Title: Does Cefoxitin or Piperacillin-Tazobactam Prevent Postoperative Surgical Site Infections After Pancreatoduodenectomy?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Indiana University (Other); Massachusetts General Hospital (Other); Thomas Jefferson University (Other); Washington University School of Medicine (Other); Advocate Illinois Masonic Medical Center (Other); Baptist Memorial Health Care Corporation (Other); Baylor Scott and White Health (Other); The Cleveland Clinic (Other); Emory University (Other); Fox Chase Cancer Center (Other); Gundersen Lutheran Medical Center (Unknown); Hackensack Meridian Health (Other); Hamilton Health Sciences Center (Unknown); Intermountain Health Care, Inc. (Other); Jersey Shore Medical Center (Hackensack Meridian) (Unknown); Johns Hopkins University (Other); Montefiore Medical Center/Albert Einstein College of Medicine (Unknown); North Shore University HealthSystem (Unknown); Milton S. Hershey Medical Center (Other); Rhode Island Hospital (Other); Stony Brook Medicine (Unknown); Sunnybrook Health Sciences Centre, Canada (Unknown); Temple University (Other); Ohio State University (Other); The Ottowa Hospital/University of Ottowa (Unknown); University of California, Davis (Other); University of Chicago (Other); University of Iowa (Other); University of Texas Southwestern Medical Center (Other); University of Utah (Other); University of Wisconsin, Madison (Other); Providence Health & Services (Other); Albany Medical College (Other); Northwestern University (Other); Universtiy of Mississippi Medical Center (Unknown); Mount Sinai Hospital, New York (Other); Brody School of Medicine at East Carolina University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-418
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; Pancreas Cancer; Pancreatic Diseases
Keywords: pancreatoduodenectomy; 17-418; cefoxitin; piperacillin-tazobactam
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases | interventions — Cefoxitin; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cefoxitin (Active Comparator)
  Interventions: Drug: Cefoxitin
- Piperacillin-tazobactam (Experimental)
  Interventions: Drug: Piperacillin-tazobactam

INTERVENTIONS:
Drug: Cefoxitin — Participants will receive one dose of cefoxitin within 1 hour of incision time, redosed every 2-4 hours in the operating room until closure of the incision, and discontinued within 24 hours after anesthesia end time.
  Arms: Cefoxitin
Drug: Piperacillin-tazobactam — Participants will receive one dose of piperacillin-tazobactam within 1 hour of incision time, redosed every 2-4 hours in the operating room until closure of the incision, and discontinued within 24 hours after anesthesia end time.
  Arms: Piperacillin-tazobactam

SUMMARY:
The purpose of this study is to figure out which commonly used antibiotic, cefoxitin or piperacillin-tazobactam, is better at decreasing the rate of surgical site infections after pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Patients undergoing elective pancreatoduodenectomy (PD) for any diagnosis/indication

Exclusion Criteria:

* Patients undergoing a minimally invasive PD, such as laparoscopic or robotic PD
* Patients with known and documented allergies to any of the penicillins, cephalosporins, or β-lactamase inhibitors
* Patients who are otherwise ineligible to receive the antibiotics in this study
* Patients highly unlikely to undergo PD according to the surgeon's judgment, such as conditions amenable to pancreas enucleation, ampullectomy, etc.
* Patients with long-term glucocorticosteroid use. The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Patients unable to provide informed consent
* Creatinine clearance (CrCl) </= 40 mL/min
* Patients receiving hemodialysis or peritoneal dialysis
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test
* Patients with a known bacterial infection present at the time of surgery or who received antimicrobial therapy within 7 days prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 967 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D'Angelica, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (32):
- United States (29):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern Medicine (Data Collection), Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Washington School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Hackensack Meridian Health / Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memoral Sloan Kettering Westchester (Consent only), Harrison, New York
  - Mount Sinai Hospital, New York, New York
  - Mount Sinai West, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Health Systems (Montefiore Medical Center), The Bronx, New York
  - Duke University, Durham, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Ohio State University, Columbus, Ohio
  - Providence Health & Services (Portland Med Ctr), Portland, Oregon
  - Pennsylvania State Hershey, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Baptist Memorial Healthcare, Memphis, Tennessee
  - Baylor Scott & White Health, Dallas, Texas
  - Intermountain Healthcare, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Canada (3):
  - Hamilton Health Sciences Center (Juravinski Hospital), Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Angelica MI, Ellis RJ, Liu JB, Brajcich BC, Gonen M, Thompson VM, Cohen ME, Seo SK, Zabor EC, Babicky ML, Bentrem DJ, Behrman SW, Bertens KA, Celinski SA, Chan CHF, Dillhoff M, Dixon MEB, Fernandez-Del Castillo C, Gholami S, House MG, Karanicolas PJ, Lavu H, Maithel SK, McAuliffe JC, Ott MJ, Reames BN, Sanford DE, Sarpel U, Scaife CL, Serrano PE, Smith T, Snyder RA, Talamonti MS, Weber SM, Yopp AC, Pitt HA, Ko CY. Piperacillin-Tazobactam Compared With Cefoxitin as Antimicrobial Prophylaxis for Pancreatoduodenectomy: A Randomized Clinical Trial. JAMA. 2023 May 9;329(18):1579-1588. doi: 10.1001/jama.2023.5728. PMID 37078771
- [Derived] Nevarez NM, Brajcich BC, Liu J, Ellis R, Ko CY, Pitt HA, D'Angelica MI, Yopp AC. Cefoxitin versus piperacillin-tazobactam as surgical antibiotic prophylaxis in patients undergoing pancreatoduodenectomy: protocol for a randomised controlled trial. BMJ Open. 2021 Mar 4;11(3):e048398. doi: 10.1136/bmjopen-2020-048398. PMID 33664081
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cefoxitin | Piperacillin-tazobactam
Started | 484 | 483
Completed | 400 | 378
Not Completed | 84 | 105
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Unresectable at surgery | 39 | 58
Not completed — Patient canceled surgery | 5 | 14
Not completed — Preoperative progression | 14 | 9
Not completed — Preoperative infection | 10 | 4
Not completed — Kidney insufficiency | 1 | 0
Not completed — Drug allergy | 0 | 2
Not completed — Operation changed to different resection | 9 | 0
Not completed — Preoperative steroid | 0 | 3
Not completed — Accrual Closed | 2 | 0
Not completed — Operation changed to different resection | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefoxitin | Piperacillin-tazobactam | Total
Number analyzed (Participants) | 400 | 378 | 778
Age, Continuous [Median (Full Range); unit: years] | 68.0 [59.8 to 73.9] | 66.8 [59.6 to 73.8] | 67.0 [59.6 to 73.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 145 | 322
  Male | 223 | 233 | 456
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 307 | 280 | 587
  Unknown or Not Reported | 87 | 92 | 179
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 19 | 46
  White | 276 | 258 | 534
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 93 | 92 | 185
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 400 | 378 | 778

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Evaluated for the Effectiveness of Cefoxitin as a Surgical Antibiotic Prophylaxis.
Description: To compare the effectiveness of cefoxitin, a second generation cephalosporin (Cohort 1), with piperacillin-tazobactam, a broad-spectrum penicillin (Cohort 2), as surgical antibiotic prophylaxis in decreasing the overall rate of postoperative SSIs in patients undergoing PD. The primary endpoint, overall SSI rate, is defined as superficial incisional SSI, deep incisional SSI, or organ/space SSI within the first 30 days after the operation, as defined according to the ACS NSQIP data collection operations manual.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cefoxitin | Piperacillin-tazobactam
Number analyzed (Participants) | 400 | 378
Participants | 400 | 378

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cefoxitin | Piperacillin-tazobactam
All-Cause Mortality (participants affected / at risk) | 10/400 | 5/378
Serious Adverse Events (participants affected / at risk) | 10/400 | 5/378
Other Adverse Events (participants affected / at risk) | 0/400 | 0/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cefoxitin (N=400) | Piperacillin-tazobactam (N=378)
Death (General disorders) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03269994/Prot_SAP_000.pdf